CLINICAL TRIAL: NCT00461045
Title: Phase 2 Clinical Trial of NPI-0052 in Patients With Relapsed or Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPI-0052-101
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; proteasome inhibitor; relapsed; refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — marizomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRZ 0.5 mg/m^2 (Experimental): Twice-weekly dosing with 2-hour IV infusions on days 1,4,8, and 11 of 3-week cycles
  Interventions: Drug: MRZ 0.5 mg/m^2

INTERVENTIONS:
Drug: MRZ 0.5 mg/m^2 — NPI-0052 0.5 mg/m2 administered IV over 2 hours on Days 1, 4, 8, and 11 in each 21-day cycle
  Other Names: Marizomib; NPI-0052

SUMMARY:
This is a Phase 2, open-label, multicenter study examining the safety, pharmacokinetics and pharmacodynamics, and best overall response to escalating doses of the proteasome inhibitor NPI-0052 (also known as marizomib) in patients with relapsed or relapsed/refractory multiple myeloma. NPI-0052 is a novel, second generation proteasome inhibitor that prevents the breakdown of proteins involved in signal transduction which blocks growth and survival in cancer cells. The study is a Phase 2 study and is a 2-stage efficacy design in a selected subgroup of patients (Arm C) treated with the recommended phase 2 dose of NPI-0052, as determined in a previously completed Phase 1 study. The study is to evaluate the safety and any preliminary evidence of efficacy of NPI-0052 in multiple myeloma patients who have previously received carfilzomib (PR-171, Kyprolis™) and subsequently had disease progression.

ELIGIBILITY:
Inclusion Criteria: Prior to Amendment 13:

* Age 18 years.
* Karnofsky Performance Status (KPS) score 70%.
* All patients must have histologic evidence of multiple myeloma. Evidence of relapsed or relapsed/refractory disease for which no other approved treatment is available and clinically indicated. In addition, patients may have undergone prior bone marrow transplantation. For patients treated at the Recommended Phase 2 Dose patients are required to have measurable relapsed or relapsed/refractory disease. Disease must be assessed within 28 days prior to treatment initiation.

  1. Measurable disease is defined as one of the following:

     * Serum M-protein ≥0.5 g/dL
     * Urine M-protein ≥200 mg/24 hours
     * Involved serum free light chain (FLC) level ≥10 mg/dL, provided the serum FLC ratio is abnormal
  2. Relapsed and Refractory are defined as:

     * Must have received at least 2 prior treatment regimens.
     * Must have received prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of bortezomib (either in separate regimens or within the same regimen).
     * Must have received a cytotoxic chemotherapy agent (eg, alkylating agent).
     * Relapsed Disease: Must have progressive disease after having achieved at least stable disease for at least one cycle of treatment during at least one prior regimen.
     * Refractory Disease: Must have documented evidence of progressive disease during or within 60 days (measured from the end of the last cycle) of completing the most recently received anti-myeloma drug regimen prior to study entry
* All AEs resulting from prior chemotherapy, surgery, or radiotherapy must have resolved to NCI-CTCAE Grade 1 (except for hematologic parameters outlined below).
* The following laboratory results, within 7 days prior to NPI-0052 administration (transfusions and/or growth factor support may be used with discretion by the Investigator during Screening):

  * Hemoglobin 8 g/dL
  * Absolute neutrophil count 0.5 × 109/L
  * Platelet count 30 × 109/L
  * Serum bilirubin 1.5 × ULN
  * AST 2.5 × ULN
  * Serum creatinine 1.5 × ULN
  * Creatinine clearance ≥40 mL/min
* Signed informed consent.
* Must have previously received at least 2 cycles of carfilzomib (as a single agent or in combination with other agents) and subsequently had disease progression during or within 60 days of carfilzomib therapy. Carfilzomib does not have to be the most recent therapy that the patient has received, but patients must have documented disease progression during or within 60 days of their last anti-myeloma therapy

Inclusion Criteria Amendment 13:

* Age 18 years.
* Karnofsky Performance Status score 70%.
* All patients must have histologic evidence of multiple myeloma and evidence of relapsed or relapsed/refractory disease as defined below Patients are required to have measurable relapsed or relapsed/refractory disease. Disease must be assessed within 28 days prior to treatment initiation.

  1. Measurable disease defined as one of the following:

     * Serum M-protein ≥0.5 g/dL
     * Urine M-protein ≥200 mg/24 hours
     * Involved serum free light chain (FLC) level ≥10 mg/dL provided the serum FLC ratio is abnormal
  2. Relapsed and Refractory are defined as:

     * Must have received at least 2 prior treatment regimens.
     * Must have received prior treatment with at least 2 cycles of an immunomodulator (lenalidomide or pomalidomide or thalidomide).
     * Must have previously received at least 2 cycles of carfilzomib (as a single agent or in combination with other agents) and subsequently had disease progression during or within 60 days of carfilzomib therapy. Carfilzomib does not have to be the most recent therapy that the patient has received, but patients must have documented disease progression during or within 60 days of their last anti-myeloma therapy. Patients may also have received bortezomib.

In addition, patients may have undergone prior cytotoxic chemotherapy, bone marrow transplantation and previously participated in other clinical trials.

* Relapsed Disease: Must have progressive disease after having achieved at least stable disease for at least one cycle of treatment during at least one prior regimen.
* Refractory Disease: Must have documented evidence of progressive disease during or within 60 days (measured from the end of the last cycle) of completing the most recently received anti-myeloma drug regimen prior to study entry.

  * All Adverse Events resulting from prior chemotherapy, surgery, or radiotherapy, must have resolved to CTCAE Grade 1 (except for hematologic parameters outlined below).
  * The following laboratory results, within 7 days of NPI-0052 administration (transfusions and/or growth factor support may be used with discretion by the Investigator during the screening period):
* Hemoglobin 8 g/dL
* Absolute neutrophil count 0.5 x 109/L
* Platelet count 30 x 109/L
* Serum bilirubin 1.5 x ULN
* AST 2.5 x ULN
* Serum creatinine 1.5 x ULN
* Creatinine clearance ≥40 mL/min -Signed informed consent.

Exclusion Criteria:

* Administration of chemotherapy, biological, immunotherapy, or investigational agent (therapeutic or diagnostic) within 14 days prior to receipt of study medication (this washout period can be reduced to 7 days for biologically targeted therapies (eg, bortezomib, carfilzomib, thalidomide, lenalidomide, pomalidomide, and dexamethasone or equivalent), provided the patient has recovered from the toxicity from these regimens per Inclusion Criterion #4). Patients must be 6 weeks from last dose of nitrosourea and 12 weeks from BMT. Patients must be 2 weeks from last dose of radiation.
* Patients with Grade >1 proteinuria (1 g/24 hour excluding M proteins = urine paraprotein subtracted from total urine protein), untreated urinary tract infection, as well as any pre existing kidney disease (acute or chronic) that in the Investigator's assessment would impose excessive risk to the patient.
* Patients with evidence of mucosal or internal bleeding and/or platelet refractory (ie, unable to maintain platelet count 30 × 109/L).
* Significant cardiac disease defined as:

  * Patients with congenital long QT syndrome;
  * Congestive heart failure of Class III or IV of the NYHA classification;
  * History of myocardial infarction or ischemia within 12 months of study enrollment.
* Abnormal left ventricular ejection fraction (LVEF) (< lower limit of normal as defined by the study site for a patient of that age) by echocardiogram (ECHO) or multiple-gated angiography (MUGA).
* Patients with a prior hypersensitivity reaction of CTCAE Grade >3 to therapy containing propylene glycol or ethanol.
* Pregnant or breast-feeding women. Female patients must be postmenopausal or surgically sterile, or they must agree to use acceptable methods of birth control (ie, a hormonal contraceptive with barrier method, intra-uterine device, diaphragm with spermicidal or condom with spermicide, or abstinence) for the duration of the study and for one month following study completion. Female patients with childbearing potential must have a negative serum pregnancy test within the 7 days before the first NPI-0052 administration. Male patients must be surgically sterile or agree to use an acceptable method of contraception.
* Active uncontrolled bacterial or fungal infection requiring systemic therapy; infection requiring parenteral antibiotics.
* Known to be HIV positive or positive and active for hepatitis A, B, or C.
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include infection requiring parenteral or oral anti-infective treatment or any altered mental status or psychiatric condition that would interfere with an understanding of the informed consent.
* Unwilling or unable to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Reich, MD, Study Director — Triphase Research and Development I Corp
Locations (6):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, School of Medicine, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Bross PF, Kane R, Farrell AT, Abraham S, Benson K, Brower ME, Bradley S, Gobburu JV, Goheer A, Lee SL, Leighton J, Liang CY, Lostritto RT, McGuinn WD, Morse DE, Rahman A, Rosario LA, Verbois SL, Williams G, Wang YC, Pazdur R. Approval summary for bortezomib for injection in the treatment of multiple myeloma. Clin Cancer Res. 2004 Jun 15;10(12 Pt 1):3954-64. doi: 10.1158/1078-0432.CCR-03-0781. No abstract available. PMID 15217925
- [Background] Chauhan D, Li G, Podar K, Hideshima T, Mitsiades C, Schlossman R, Munshi N, Richardson P, Cotter FE, Anderson KC. Targeting mitochondria to overcome conventional and bortezomib/proteasome inhibitor PS-341 resistance in multiple myeloma (MM) cells. Blood. 2004 Oct 15;104(8):2458-66. doi: 10.1182/blood-2004-02-0547. Epub 2004 Jun 24. PMID 15217830
- [Background] Chauhan D, Li G, Shringarpure R, Podar K, Ohtake Y, Hideshima T, Anderson KC. Blockade of Hsp27 overcomes Bortezomib/proteasome inhibitor PS-341 resistance in lymphoma cells. Cancer Res. 2003 Oct 1;63(19):6174-7. PMID 14559800
- [Background] Chauhan D, Catley L, Li G, Podar K, Hideshima T, Velankar M, Mitsiades C, Mitsiades N, Yasui H, Letai A, Ovaa H, Berkers C, Nicholson B, Chao TH, Neuteboom ST, Richardson P, Palladino MA, Anderson KC. A novel orally active proteasome inhibitor induces apoptosis in multiple myeloma cells with mechanisms distinct from Bortezomib. Cancer Cell. 2005 Nov;8(5):407-19. doi: 10.1016/j.ccr.2005.10.013. PMID 16286248
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- [Background] Cheson BD, Pfistner B, Juweid ME, et al. Revised Response Criteria for Malignant Lymphomas. From the Members of the International Harmonization Project (IHP) of the Competence Network Malignant Lymphoma, 47th Annual Meeting of the American Society of Hematology. Blood. 2005 Nov;106: abstract #18
- [Background] ClinicalTrials.gov. Phase 3 Study With Carfilzomib and Dexamethasone Versus Velcade and Dexamethasone for Relapsed Multiple Myeloma Patients (ENDEAVOR). ClinicalTrials.gov Identifier: NCT01568866.
- [Background] DeGeorge JJ, Ahn CH, Andrews PA, Brower ME, Giorgio DW, Goheer MA, Lee-Ham DY, McGuinn WD, Schmidt W, Sun CJ, Tripathi SC. Regulatory considerations for preclinical development of anticancer drugs. Cancer Chemother Pharmacol. 1998;41(3):173-85. doi: 10.1007/s002800050726. PMID 9443633
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Dy GK, Thomas JP, Wilding G, Bruzek L, Mandrekar S, Erlichman C, Alberti D, Binger K, Pitot HC, Alberts SR, Hanson LJ, Marnocha R, Tutsch K, Kaufmann SH, Adjei AA. A phase I and pharmacologic trial of two schedules of the proteasome inhibitor, PS-341 (bortezomib, velcade), in patients with advanced cancer. Clin Cancer Res. 2005 May 1;11(9):3410-6. doi: 10.1158/1078-0432.CCR-04-2068. PMID 15867242
- [Background] 12. Facon T, Dimopoulos M, Dispenzieri A, et al. Initial Phase 3 Results Of The First (Frontline Investigation Of Lenalidomide + Dexamethasone Versus Standard Thalidomide) Trial (MM-020/IFM 07 01) In Newly Diagnosed Multiple Myeloma (NDMM) Patients (Pts) Ineligible For Stem Cell Transplantation (SCT). 2013; ASH Annual Meeting Plenary Session, Sunday, December 8, 2013: 2:55 PM
- [Background] Feling RH, Buchanan GO, Mincer TJ, Kauffman CA, Jensen PR, Fenical W. Salinosporamide A: a highly cytotoxic proteasome inhibitor from a novel microbial source, a marine bacterium of the new genus salinospora. Angew Chem Int Ed Engl. 2003 Jan 20;42(3):355-7. doi: 10.1002/anie.200390115. No abstract available. PMID 12548698
- [Background] Fleming TR. One-sample multiple testing procedure for phase II clinical trials. Biometrics. 1982 Mar;38(1):143-51. PMID 7082756
- [Background] Goy A, Younes A, McLaughlin P, Pro B, Romaguera JE, Hagemeister F, Fayad L, Dang NH, Samaniego F, Wang M, Broglio K, Samuels B, Gilles F, Sarris AH, Hart S, Trehu E, Schenkein D, Cabanillas F, Rodriguez AM. Phase II study of proteasome inhibitor bortezomib in relapsed or refractory B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2005 Feb 1;23(4):667-75. doi: 10.1200/JCO.2005.03.108. Epub 2004 Dec 21. PMID 15613697
- [Background] Hamilton AL, Eder JP, Pavlick AC, Clark JW, Liebes L, Garcia-Carbonero R, Chachoua A, Ryan DP, Soma V, Farrell K, Kinchla N, Boyden J, Yee H, Zeleniuch-Jacquotte A, Wright J, Elliott P, Adams J, Muggia FM. Proteasome inhibition with bortezomib (PS-341): a phase I study with pharmacodynamic end points using a day 1 and day 4 schedule in a 14-day cycle. J Clin Oncol. 2005 Sep 1;23(25):6107-16. doi: 10.1200/JCO.2005.01.136. PMID 16135477
- [Background] Kisselev AF, Goldberg AL. Proteasome inhibitors: from research tools to drug candidates. Chem Biol. 2001 Aug;8(8):739-58. doi: 10.1016/s1074-5521(01)00056-4. PMID 11514224
- [Background] Kondagunta GV, Drucker B, Schwartz L, Bacik J, Marion S, Russo P, Mazumdar M, Motzer RJ. Phase II trial of bortezomib for patients with advanced renal cell carcinoma. J Clin Oncol. 2004 Sep 15;22(18):3720-5. doi: 10.1200/JCO.2004.10.155. PMID 15365068
- [Background] KYPROLIS™ (carfilzomib) for Injection Prescribing Information. Onyx Pharmaceuticals, Inc., South San Francisco, CA; 07/2012. http://www.kyprolis.com/Areas/Hcp/content/pdfs/PI.pdf
- [Background] Macherla VR, Mitchell SS, Manam RR, Reed KA, Chao TH, Nicholson B, Deyanat-Yazdi G, Mai B, Jensen PR, Fenical WF, Neuteboom ST, Lam KS, Palladino MA, Potts BC. Structure-activity relationship studies of salinosporamide A (NPI-0052), a novel marine derived proteasome inhibitor. J Med Chem. 2005 Jun 2;48(11):3684-7. doi: 10.1021/jm048995+. PMID 15916417
- [Background] Anderson KC, Alsina M, Bensinger W, Biermann JS, Chanan-Khan A, Cohen AD, Devine S, Djulbegovic B, Gasparetto C, Huff CA, Jagasia M, Medeiros BC, Meredith R, Raje N, Schriber J, Singhal S, Somlo G, Stockerl-Goldstein K, Tricot G, Vose JM, Weber D, Yahalom J, Yunus F; National Comprehensive Cancer Network. NCCN clinical practice guidelines in oncology: multiple myeloma. J Natl Compr Canc Netw. 2009 Oct;7(9):908-42. doi: 10.6004/jnccn.2009.0061. No abstract available. PMID 19878637
- [Background] National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology. http://www.nccn.org/professionals/physician_gls/pdf/myeloma.pdf. Multiple Myeloma (Version 2.2013). Accessed 29 August 2013
- [Background] O'Connor OA, Wright J, Moskowitz C, Muzzy J, MacGregor-Cortelli B, Stubblefield M, Straus D, Portlock C, Hamlin P, Choi E, Dumetrescu O, Esseltine D, Trehu E, Adams J, Schenkein D, Zelenetz AD. Phase II clinical experience with the novel proteasome inhibitor bortezomib in patients with indolent non-Hodgkin's lymphoma and mantle cell lymphoma. J Clin Oncol. 2005 Feb 1;23(4):676-84. doi: 10.1200/JCO.2005.02.050. Epub 2004 Dec 21. PMID 15613699
- [Background] Palumbo A, Mina R. Management of older adults with multiple myeloma. Blood Rev. 2013 May;27(3):133-42. doi: 10.1016/j.blre.2013.04.001. Epub 2013 Apr 25. PMID 23623929
- [Background] Penta JS, Rozencweig M, Guarino AM, Muggia FM. Mouse and large-animal toxicology studies of twelve antitumor agents: relevance to starting dose for phase I clinical trials. Cancer Chemother Pharmacol. 1979;3(2):97-101. doi: 10.1007/BF00254979. No abstract available. PMID 116778
- [Background] Pfistner B, Diehl V, Greb A, Cheson B. International harmonization of trial parameters in malignant lymphoma. Eur J Haematol Suppl. 2005 Jul;(66):53-4. doi: 10.1111/j.1600-0609.2005.00455.x. PMID 16007869
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775
- [Background] Richardson PG, Sonneveld P, Schuster MW, Irwin D, Stadtmauer EA, Facon T, Harousseau JL, Ben-Yehuda D, Lonial S, Goldschmidt H, Reece D, San-Miguel JF, Blade J, Boccadoro M, Cavenagh J, Dalton WS, Boral AL, Esseltine DL, Porter JB, Schenkein D, Anderson KC; Assessment of Proteasome Inhibition for Extending Remissions (APEX) Investigators. Bortezomib or high-dose dexamethasone for relapsed multiple myeloma. N Engl J Med. 2005 Jun 16;352(24):2487-98. doi: 10.1056/NEJMoa043445. PMID 15958804
- [Background] Ruiz S, Krupnik Y, Keating M, Chandra J, Palladino M, McConkey D. The proteasome inhibitor NPI-0052 is a more effective inducer of apoptosis than bortezomib in lymphocytes from patients with chronic lymphocytic leukemia. Mol Cancer Ther. 2006 Jul;5(7):1836-43. doi: 10.1158/1535-7163.MCT-06-0066. PMID 16891470
- [Background] Siegel DS, Martin T, Wang M, Vij R, Jakubowiak AJ, Lonial S, Trudel S, Kukreti V, Bahlis N, Alsina M, Chanan-Khan A, Buadi F, Reu FJ, Somlo G, Zonder J, Song K, Stewart AK, Stadtmauer E, Kunkel L, Wear S, Wong AF, Orlowski RZ, Jagannath S. A phase 2 study of single-agent carfilzomib (PX-171-003-A1) in patients with relapsed and refractory multiple myeloma. Blood. 2012 Oct 4;120(14):2817-25. doi: 10.1182/blood-2012-05-425934. Epub 2012 Jul 25. PMID 22833546
- [Background] Simon R, Freidlin B, Rubinstein L, Arbuck SG, Collins J, Christian MC. Accelerated titration designs for phase I clinical trials in oncology. J Natl Cancer Inst. 1997 Aug 6;89(15):1138-47. doi: 10.1093/jnci/89.15.1138. PMID 9262252
- [Background] Suzuki E, Jazirehi A, Palladino M, Bonavida B. Chemosensitization of Drug and Rituximab Resistant Daudi B-NHL Clones to Drug-Induced Apoptosis by the Proteasome Inhibitor NPI-0052. 47th Annual Meeting of the American Society for Hematology. Blood. 2005;106: abstract #1521
- [Background] Yasui H, Hideshima T, Hamasaki M, Roccaro AM, Shiraishi N, Kumar S, Tassone P, Ishitsuka K, Raje N, Tai YT, Podar K, Chauhan D, Leoni LM, Kanekal S, Elliott G, Munshi NC, Anderson KC. SDX-101, the R-enantiomer of etodolac, induces cytotoxicity, overcomes drug resistance, and enhances the activity of dexamethasone in multiple myeloma. Blood. 2005 Jul 15;106(2):706-12. doi: 10.1182/blood-2005-02-0838. Epub 2005 Mar 31. PMID 15802527
- [Derived] Richardson PG, Zimmerman TM, Hofmeister CC, Talpaz M, Chanan-Khan AA, Kaufman JL, Laubach JP, Chauhan D, Jakubowiak AJ, Reich S, Trikha M, Anderson KC. Phase 1 study of marizomib in relapsed or relapsed and refractory multiple myeloma: NPI-0052-101 Part 1. Blood. 2016 Jun 2;127(22):2693-700. doi: 10.1182/blood-2015-12-686378. Epub 2016 Mar 23. PMID 27009059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRZ 0.5 mg/m^2
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Baseline Height [Mean (Standard Deviation); unit: cm] | 170.97 (12.152)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 77.27 (17.825)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.893 (0.2629)
Fertility Status [Count of Participants; unit: Participants]
  Potential able to bear children | 0
  Surgically sterile | 1
  Post menopausal | 4
  Male | 10
Karnofsky Performance Status (KPS) Score [Mean (Full Range); unit: KPS Score] — KPS Score: 100=Normal, no complaints; 90=Able to carry on normal activity, minor signs or symptoms of disease; 80=Normal activity with effort; 70= Unable to carry on normal activity or perform active work, cares for self.
  KPS Score | 87.3 [70.0 to 100.0]
Time Since Initial Diagnosis [Mean (Standard Deviation); unit: years] | 5.2 (3.79)
Number of Relapses [Number; unit: participants]
  1 Relapse | 0
  2 Relapses | 2
  3 Relapses | 2
  >3 Relapses | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Exhibiting a Given Overall Response as Determined by Investigator
Description: Disease response and progression were determined by the investigator using the International Myeloma Working Group Uniform Response Criteria (IMWG-URC). Overall response rate includes patients with a best response of PR of better. Stringent complete response (CR) includes immunophenotypic CR and molecular CR in addition to stringent CR.
Time Frame: Through study completion, an average of 6.09 weeks.
Measure: Number; unit: participants
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 15
participants
  Stringent Complete Response (sCR) or better | 0
  Complete Response (CR) | 0
  Very Good Partial Response (VGPR) | 0
  Partial Response (PR) | 0
  Minimal Response (MR) | 0
  Stable Disease (SD) | 4
  Progressive Disease (PD) | 9
  Not Evaluated | 2

2. Secondary Outcome: Duration of MRZ Treatment
Description: Duration of treatment is defined as the last dose date minus the first dose date of the dose cohort plus 1 expressed in weeks.
Time Frame: Through study completion, an average of 6.09 weeks.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 15
weeks | 6.09 (4.661)

3. Secondary Outcome: Number of Cycles of Marizomib (MRZ)
Time Frame: Through study completion, an average of 6.09 weeks.
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 15
cycles | 2.6 (1.45)

4. Secondary Outcome: Number of Patients Receiving Marizomib (MRZ) in Each Cycle
Description: A patient was counted in a cycle if the patient received at least one dose of study drug during the cycle.
Time Frame: Through study completion, an average of 6.09 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 15
Participants
  Cycle 1 | 15
  Cycle 2 | 12
  Cycle 3 | 6
  Cycle 4 | 3
  Cycle 5 | 2
  Cycle 6 | 1

5. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events were graded using NCI-CTCAE (version 4.3). TEAEs are defined as any adverse event with an onset date between the date of first dose and 30 days after the date of last dose of any study drug.
  Treatment-related adverse events are adverse events considered related to at least one study drug by the investigator (NPI-002, dexamethasone), including those with unknown relationship.
Time Frame: Through study completion, an average of 6.09 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 15
Participants
  At least one TEAE | 15
  At least one treatment related TEAE | 14
  At least one NPI-0052 related TEAE | 13
  At least one grade ≥3 TEAE | 12
  At least one treatment related grade ≥3 TEAE | 8
  At least one NPI-0052 related grade ≥3 TEAE | 5
  At least one serious TEAE | 7
  At least one treatment related serious TEAE | 4
  At least one NPI-0052 related serious TEAE | 1

6. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: as for outcome 5
Time Frame: Through study completion, an average of 6.09 weeks.
Measure: Number; unit: TEAEs
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 15
TEAEs
  Number of TEAEs | 149
  Number of treatment related TEAEs | 73
  Number of NPI-0052 related TEAEs | 50
  Number of grade ≥3 TEAEs | 41
  Number of treatment related grade ≥3 TEAEs | 16
  Number of NPI-0052 realted grade ≥3 TEAEs | 9
  Number of serious TEAEs | 21
  Number of treatment related serious TEAEs | 5
  Number of NPI-0052 related serious TEAEs | 1

7. Secondary Outcome: Maximum Observed Blood Drug Concentration (Cmax)
Time Frame: Samples collected on Cycle 1 Day 1 and Cycle 1 Day 11.
Population: The sponsor elected not to analyze the pharmacokinetic (PK) samples collected, therefore, no PK results are obtained.
Arm/Group | MRZ 0.5 mg/m^2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | MRZ 0.5 mg/m^2
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRZ 0.5 mg/m^2 (N=15)
Sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Renal failure acute (Renal and urinary disorders) | 2
Cardiac Failure Congestive (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Adverse Drug Reaction (General disorders) | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 1
Arthritis Bacterial (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Endocarditis Bacterial (Infections and infestations) | 1
Escherichia Bacteraemia (Infections and infestations) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1
Embolic Stroke (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRZ 0.5 mg/m^2 (N=15)
Fatigue (General disorders) | 9
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Gait disturbance (General disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Hallucination, Visual (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Tenderness (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Adverse Drug Reaction (General disorders) | 1
Infusion Site Erythema (General disorders) | 1
Vessel Puncture Site Pain (General disorders) | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 2
Arthritis Bacterial (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Endocarditis Bacterial (Infections and infestations) | 1
Escherichia Bacteraemia (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1
Blood Creatinine Increased (Investigations) | 2
Weight Decreased (Investigations) | 2
International Normalised Ratio Increased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 1
Platelet Count Decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Metabolic Alkalosis (Metabolism and nutrition disorders) | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 2
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Aphasia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Embolic Stroke (Nervous system disorders) | 1
Head Discomfort (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 5
Confusional State (Psychiatric disorders) | 2
Dysphoria (Psychiatric disorders) | 1
Pressure of Speech (Psychiatric disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Skin Mass (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No